CLINICAL TRIAL: NCT05405296
Title: Performance Evaluation of the Molbio Diagnostics Truenat™MTB Plus/COVID-19for TB and COVID-19case Detection Using Prospectively Collected NP (Nasopharyngeal) Swabs and Sputum Samples From Participants With Symptoms Suggestive of TB
Brief Title: Evaluation of the Truenat™MTB Plus/COVID-19 Test for TB (Tuberculosis) and COVID-19 (SARS-CoV2)
Acronym: Truenat COMBO
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: TB050
Record Dates: First submitted 2022-06-03; First posted 2022-06-06 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: TB; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tongue swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Truenat™ MTB Plus/COVID-19 — Truenat™ MTB Plus/COVID-19is a disposable, room temperature stable, chip-based Real Time duplex PCR test, along with freeze dried PCR reagents provided in microtube for performing Real Time PCR for infectious disease and runs on the Truelab® Real Time micro-PCR Analyzer.

SUMMARY:
This is a prospective, multicentre study in which the accuracy of the Molbio Diagnostics Truenat™ MTB (Mycobacterium tuberculosis) Plus/COVID-19multiplex will be assessed for TB and COVID-19 case detection using prospectively collected NP swabs and sputum samples from patients with symptoms suggestive of TB.

The overall study period is of 24 months which includes telephonic follow-up of the baseline COVID-19negative patients at 2 weeks and of all participants at 2 months.

DETAILED DESCRIPTION:
Adult patient with presumptive TB will be screened for inclusion at 4 geographically diverse participating centres in high TB burden countries. This will be the first large scale evaluation on prospectively collected fresh samples.

Telephonic follow-up visits at 2 weeks (for baseline COVID-19 negative patients) and 2 months (for all participants) after enrolment will help overcome the challenges of using MRS only. Follow-up will be conducted telephonically two weeks post-enrolment for participants who tested negative for COVID-19at enrolment to determine any change in status -this is intended to account for participants who may have tested 'early' for COVID-19at enrolment (false negative) but subsequently developed symptoms or tested COVID-19positive. Similarly, investigators will conduct a telephonic follow-up two months post-enrolment among all participants to determine if: 1) participants diagnosed with confirmed TB at enrolment were linked to treatment; and 2) assess if any new TB diagnoses were made.

This multi-center study will evaluate the performance of the Truenat™ MTB (Mycobacterium tuberculosis) Plus/COVID-19multiplex test using prospectively collected NP swabs and sputum samples from patients with symptoms suggestive of TB and collect alternative tongue swab samples for further research use. The data gathered from this study, will form part of the dossier to be submitted to WHO (world health organization) for review.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years); and
* Able to provide written informed consent in their chosen language; and
* Self-report at least one or more symptoms suggestive of pulmonary TB*; and
* Willing to return for a day 2 visit
* Willing to provide oral swab samples for biobanking * cough ≥2 weeks, fever, night sweats or unintended weight-loss

Exclusion Criteria:

* Any tuberculosis preventive therapy (TPT) within 6 months prior to enrolment
* Any anti-TB treatment within 60 days prior to enrolment (not current episode)
* Unable to provide 3ml of sputum, nasopharyngeal and tongue swabs on Day1
* Unable to provide all study samples before starting the 3rddose of anti-TB treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study focuses on adults with presumptive TB. Study sites are selected to maximize the generalizability of evidence generated based on the following criteria: 1) TB incidence ≥100 per 100,000 population; 2) HIV prevalence; 3) ongoing community transmission of COVID-19; and 4) laboratory and clinical study infrastructure to support participant recruitment.
  Location: the study will take place in 4different countries: South Africa, Uganda, Peru, India Prospective approval of protocol deviations to recruitment and enrolment criteria, also known as protocol waivers or exemptions, are not permitted.
Sampling Method: Probability Sample
Enrollment: 1480 (Estimated)
Dates: Start 2022-08-30 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Point estimates of sensitivity and specificity of Truenat™ MTB Plus/COVID-19 | 2 days
  Point estimates of sensitivity and specificity of Truenat™ MTB Plus/COVID-19, with 95% confidence intervals, using the defined TB MRS

SECONDARY OUTCOMES:
Point estimates of sensitivity and specificity of Truenat™ MTB Plus/COVID-19, with 95% confidence intervals, using a country-approved RT-PCR COVID-19 | 2 days
  Point estimates of sensitivity and specificity of Truenat™ MTB Plus/COVID-19, with 95% confidence intervals, using a country-approved RT-PCR ( real time polymerase chain reaction) COVID-19
Point estimates of sensitivity and specificity of Truenat™ MTB Plus/COVID-19multiplex for TB detection compared to Xpert Ultra among presumptive TB patients using a MRS | 2 days
  Point estimates of sensitivity and specificity of Truenat™ MTB Plus/COVID-19multiplex for TB detection compared to Xpert Ultra among presumptive TB patients using a MRS
Estimate of the proportion of presumptive TB patients with COVID-19 | 2 days
  Estimate of the proportion of presumptive TB patients with COVID-19 confirmed by country-approved RT-PCR Covid-19 assay) (expressed as a percentage)
Estimate of the proportion of TB patients (confirmed by MRS) with COVID-19 | 2 days
  Estimate of the proportion of TB patients (confirmed by MRS) with COVID-19(confirmed by country-approved RT-PCR Covid-19 assay) (expressed as a percentage)
Analysis of survey responses using proportions and Linkert scale averages | 2 days
  Analysis of survey responses using proportions and Linkert scale averages

CONTACTS AND LOCATIONS:
Locations (1):
- Makarere University, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Inbaraj LR, Daniel J, Sathya Narayanan MK, Srinivasalu VA, Bhaskar A, Scandrett K, Rajendran P, Kirubakaran R, Shewade HD, Malaisamy M, Padmapriyadarsini C, Takwoingi Y. Truenat MTB assays for pulmonary tuberculosis and rifampicin resistance in adults and adolescents. Cochrane Database Syst Rev. 2025 Mar 24;3(3):CD015543. doi: 10.1002/14651858.CD015543.pub2. PMID 40122135